CLINICAL TRIAL: NCT01526070
Title: Bimonthly VEGF Trap-Eye Compared to As-needed Administration or Standard Therapy for Exudative Age-Related Macular Degeneration
Brief Title: Study of Bimonthly VEGF Trap-Eye Compared to As-needed Administration or Other Therapy for Exudative Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Theodore Leng, Clinical Assistant Professor of Ophthalmology, Stanford University
Other Study IDs: SU-02012012-9068
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Exudative Age-related Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Exudative Age-Related Macular Degeneration: Patients with eAMD who received intravitreal thearpy
  Interventions: Drug: Intravitreal injection of Aflibercept

INTERVENTIONS:
Drug: Intravitreal injection of Aflibercept

SUMMARY:
Over the last several years, the standard of care for wet macular degeneration has become treatment with intravitreal injections of ranibizumab (Lucentis, Genentech), administered as frequently as every 4 weeks. In contrast, clinical trials of a soluble VEGF receptor, Aflibercept/VEGF Trap-Eye (Eylea, Regeneron Pharmaceuticals) have demonstrated maintained anatomic and visual improvement with many fewer injections (typically monthly injections for 3 months, followed by every-other-month injections, and as few as 5 injections a year). The purpose of this study is to determine whether patients who have switched from ranibizumab to VEGF Trap-Eye have comparable results.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than the age of 50 determined by a retinal physician at the Byers Eye Institute at Stanford to have exudative AMD requiring treatment.
2. Patients with an established diagnosis of exudative AMD who have been maintained on a regimen of intravitreal ranibizumab injections.
3. Postmenopausal or negative pregnancy test
4. Patients with an established diagnois of exidative AMD who have been switched from intravitreal ranibizumab to intravitreal VEGF Trap-EYE.

Exclusion Criteria:

1. Patients with any previous or concurrent history of treatment of other retinal diseases with pharmacologic agents other than ranibizumab, including verteporfin photodynamic therapy, bevacizumab, triamcinolone, or dexamethasone.
2. Patients with prior history of vitrectomy surgery in the study eye.
3. Patients enrolled in any previous or current clinical trial or study of any medication for AMD or any other retinal vascular disease, including diabetic retinopathy or retinal vein occlusion.
4. Ocular media opacity precluding proper retinal imaging
5. Inadequate pupillary dilation to achieve proper retinal imaging
6. Concurrent use of systemic anti-VEGF agents
7. CNV due to other causes, including histoplasmosis, uveitis, trauma, or myopia
8. Active or recent (< 4 weeks) or recurrent inflammation in the eye
9. Current vitreous hemorrhage in the study eye limiting visualization of the fundus
10. Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis
11. Untreated glaucoma with IOP > 25 in the eye
12. Other ocular diseases that can compromise the visual acuity of the study eye such as amblyopia and anterior ischemic optic neuropathy
13. Pregnancy or lactation
14. History of other disease, exam finding, or clinical laboratory that contraindicates the use the drug
15. Current treatment for active systemic infection
16. Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, pulmonary, renal, hepatic, endocrine, or GI disorders
17. History of recurrent significant infections or bacterial infections
18. Inability to comply with study or follow-up procedure

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with exudative age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Byers Eye Institute at Stanford, Palo Alto, California, United States